CLINICAL TRIAL: NCT07092111
Title: Efficacy of Auricular Acupuncture Therapy Via the Seirin Pyonex Needles in the Prevention of Chemotherapy-Induced Peripheral Neuropathy(CIPN) in Breast Cancer
Brief Title: Efficacy of Auricular Acupuncture Therapy in the Prevention of CIPN in Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACAA 01
Record Dates: First submitted 2025-07-02; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer
Keywords: chemotherapy-induced peripheral neuropathy; auricular acupuncture; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupuncture treatment group (Experimental): On the basis of conventional nursing, patients are treated with bilateral auricular acupuncture points (Seirin Pyonex Needles φ 0.2 mm × 1.2 mm) before chemotherapy.
  Specific operation: 1 treatment before each chemotherapy treatment, and 2 treatments a week in the 2nd and 3rd weeks of the chemotherapy interval. The patient was instructed to press the acupuncture point for 3 times/d, the pressure time was 5min, and the local swelling pain was tolerated by the patient. The doctor took the needle out for the patient after leaving it for 3 days. Treatment was continued for 4 cycles of chemotherapy, followed up for 2 months after treatment completion, and routine care was carried out during treatment.
  Interventions: Device: Auricular acupuncture treatment
- Sham acupuncture group (Sham Comparator): The treatment regimen is the same as that of the auricular acupuncture treatment group, but with a sham acupuncture (Seirin Pyonex Needles).
  Interventions: Device: Sham acupuncture group

INTERVENTIONS:
Device: Auricular acupuncture treatment — Auricular acupuncture is an innovative intradermal acupuncture, which can directly use the meridian system of the ear skin to directly transmit the received stimulation to the lesion. Its stimulation time is long, and the amount of stimulation is strong. Studies have shown that needle pricking continuously delivers an adequate dose of acupuncture stimulation by continuously stimulating Aβ, Aδ, and/or C afferent fibers from the skin and transmitting them to the brain nucleus through the ventrolateral cord of the spinal cord. It is also believed that by stimulating the cranial nerves, especially the auricular branch of the vagus nerve, the effect of sensory afferent peripheral stimulation can be enhanced, and the analgesic effect of the auricular acupoints can be achieved.
  Arms: Auricular acupuncture treatment group
Device: Sham acupuncture group — The treatment regimen is the same as that of the auricular acupuncture treatment group, but with a sham acupuncture (Seirin Pyonex Needles).
  Arms: Sham acupuncture group

SUMMARY:
Evaluate the Efficacy of Auricular Acupuncture Therapy via the Seirin Pyonex Needles in the Prevention of Chemotherapy-Induced Peripheral Neuropathy in Breast Cancer

DETAILED DESCRIPTION:
This is a Phase II Randomised Controlled Clinical Trial to evaluate the efficacy of auricular acupuncture therapy via the Seirin Pyonex Needles in the prevention of chemotherapy-induced peripheral neuropathy in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer diagnosed with stage I-III;
* Planned to receive 4 cycles of taxane chemotherapy and have not taken neurostable drugs within three months;
* 18 years old≤ age≤ 75 years old, female;
* Subjects voluntarily participate in this trial and sign the informed consent form.

Exclusion Criteria:

* Patients who have had acupuncture treatment in the past;
* After examination by a doctor, there is a local infection at or near the acupuncture site, which is not suitable for acupuncture.
* Platelets< 50,000/μL;
* Patients with CIPN≥1 grade 1 (NCI-CTCAE);
* Peripheral neuropathy or other neuropathic pain caused by diabetes mellitus or other factors related to HIV infection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient is an adult female ≥ 18 years old at the time of informed consent.
Enrollment: 110 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of CIPN at the end of the 4th chemotherapy | From date of randomization until the date of he fourth application of taxane chemotherapy (up to 12 weeks)
  Incidence of CIPN at the end of the 4th application of taxane chemotherapy (according to NCI-CTCAE V5.0)

SECONDARY OUTCOMES:
Incidence of CIPN at the end of the 3rd chemotherapy | From date of randomization until the date of he fourth application of taxane chemotherapy (up to 12 weeks)
  Incidence of CIPN before the first treatment, at the end of the first three taxane chemotherapy treatments, and at 2 months of follow-up.
CIPN neurotoxicity change | From date of randomization until the date of he fourth application of taxane chemotherapy (up to 12 weeks)
  The FACT/GOG-Ntx scale was used to evaluate the change in CIPN neurotoxicity symptom scores before the first treatment, at the end of the second taxane chemotherapy, at the end of the fourth taxane chemotherapy, and at 2 months of follow-up.
The degree of sensory impairment | From date of randomization until the date of he fourth application of taxane chemotherapy (up to 12 weeks)
  The degree of sensory impairment was assessed by Semmes-Weinstein monofilament tactile test before the first treatment, at the end of the fourth taxane chemotherapy, and at 2 months of follow-up.
The pain intensity score | From date of randomization until the date of he fourth application of taxane chemotherapy (up to 12 weeks)
  The NRS scale assessed the pain intensity score before the first treatment, at the end of the second taxane chemotherapy, at the end of the fourth taxane chemotherapy, and at 2 months of follow-up.
The General Hospital Anxiety/Depression (HAD) | From date of randomization until the date of he fourth application of taxane chemotherapy (up to 12 weeks)
  The General Hospital Anxiety/Depression (HAD) Mood Measurement Form was used to evaluate the physical fitness score of patients before the first treatment and at the end of the fourth taxane chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code